CLINICAL TRIAL: NCT05043506
Title: European Treatment Patterns and Outcomes Associated With First-Line CDK4/6 Inhibition and Hormonal Therapies Assessed in a Real-World Non-Interventional Study (EUCHARIS)
Brief Title: European Treatment Patterns and Outcomes Associated With First-Line CDK4/6 Inhibition and Hormonal Therapies
Acronym: EUCHARIS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481170; EUCHARIS (Other: Alias Study Number)
Record Dates: First submitted 2021-09-07; First posted 2021-09-14 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; Palbociclib; Real-world data; CDK4/6; effectiveness
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Aromatase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Palbociclib + aromatase inhibitor: Adult patients with advanced breast cancer patients who initiated Palbociclib + an aromatase inhibitor as first line therapy between September 1, 2016, and July 31, 2020.
  Interventions: Drug: Palbociclib + aromatase inhibitor
- Aromatase inhibitor: Adult patients with advanced breast cancer patients who initiated an aromatase inhibitor as first line therapy between January 1, 2010,, and July 31, 2020
  Interventions: Drug: Aromatase inhibitor

INTERVENTIONS:
Drug: Palbociclib + aromatase inhibitor — Palbociclib + an aromatase inhibitor therapy
  Other Names: Palbociclib + an aromatase inhibitor therapy
  Groups: Palbociclib + aromatase inhibitor
Drug: Aromatase inhibitor — Aromatase inhibitor monotherapy
  Other Names: Aromatase inhibitor monotherapy
  Groups: Aromatase inhibitor

SUMMARY:
A retrospective observational analysis of de-identified data from a multinational medical record review to describe patient characteristics, treatment patterns, and effectiveness of palbociclib + AI as first-line therapy among adult patients with HR+/HER2- advanced breast cancer (ABC) in Europe

ELIGIBILITY:
Inclusion Criteria:

* Is male or female
* Has histologically or cytologically confirmed breast cancer diagnosis (HR+/HER2- breast cancer)
* Has received a diagnosis of locally advanced breast cancer not amenable to curative radiation or surgical cure or of metastatic breast cancer (i.e., advanced breast cancer [ABC]); diagnosis may be de novo (initial diagnosis at ABC stage) or recurrent from earlier-stage disease (initial diagnosis of earlier-stage disease with subsequent progression to advanced disease)
* Has initiated a required first-line therapy of interest: Palbociclib plus AI as first-line therapy for ABC between September 1, 2016, and July 31, 2020, or AI monotherapy as first-line therapy for ABC between January 1, 2010,, and July 31, 2020
* Was aged 18 years or older at the time of diagnosis of ABC
* Is living or deceased at the time of record abstraction
* Has a complete medical record, covering treatment for ABC, including any transfer record from other facilities (if applicable) that is available to the abstractor for data abstraction

Exclusion Criteria:

* The patient's first treatment after ABC diagnosis was chemotherapy (including induction chemotherapy)
* The patient has evidence of other active malignant neoplasms within 3 years (except nonmelanoma skin cancer or carcinoma in situ) prior to diagnosis of ABC; patients diagnosed with second primary cancer after ABC diagnosis will not be excluded
* The patient has evidence of prior treatment with any CDK4/6 inhibitor (i.e. palbociclib, abemaciclib, ribociclib) in the early-stage breast cancer setting or treatment with abemaciclib or ribociclib in the ABC setting
* The patient has participated in a clinical trial related to treatment of ABC (including after first-line therapy [i.e., palbociclib plus AI or AI monotherapy])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with HR+/HER2- advanced breast cancer treated with palbociclib + an aromatase inhibitor or an aromatase inhibitor alone between January 1, 2010 to July 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 1939 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Real-world progression free survival | Time from treatment line start date to clinician assessed date of disease progression, date of death, or date of censoring
  Total time from the treatment line start date to the date of disease progression confirmed by clinician assessment or the date of censoring, as measured in months

SECONDARY OUTCOMES:
Overall survival | Time from treatment line start date to clinician assessed date of death, or date of censoring
  Time from the treatment line start to the date of confirmed death, or the date of censoring
Time to first objective tumor response | Time from treatment line start date to clinician-assessed first date of objective response or date of censoring
  Time from the date of treatment line start to the first date of clinician-assessed objective response, or the date of censoring, measured in months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (64):
- Austria (4):
  - Sankt Josef Hospital Braunau, Braunau am Inn
  - Landesklinikum Krems, Krems
  - Universitaetsklinikum Sankt Poelten, Sankt Pölten
  - Priv. Doz. OA Dr. Michael Hubalek, Schwaz
- UZ Leuven, Leuven, Belgium
- Germany (16):
  - Universitätsklinikum Würzburg Frauenklinik und Poliklinik, Würzburg, Bavaria
  - MediOnko-Institut GbR, Berlin, Brandenburg
  - Kreisklinikum Böblingen gGmbH, Frauenklinik Böblingen, Sindelfingen, Landkreis Boblingen
  - Universitatsklinikum Essen, Essen, North Rhine-Westphalia
  - Ruppiner Kliniken GmbH, Neuruppin, Ostprignitz-ruppin
  - Frauenarztpraxis, Ilsede, Peine
  - Institut für Versorgungsforschung GbR, Mainz, Rhineland-Palatinate
  - Universität des Saarlandes, Saarbrücken, Saarland
  - Studienzentrum UnterEms, Emden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Group practice Goehler, Dresden
  - Bethanien Center for Hematology and Oncology, Frankfurt
  - Überörtliche Gemeinschaftspraxis, Hamburg
  - St. Vincenz-Krankenhaus GmbH, Paderborn
  - Gynäkologie Kompetenzzentrum Praxis Dr. med. Carsten Hielscher, Stralsund
  - Medizinische Studiengesellschaft NORD-WEST GmbH, Westerstede
- Spain (20):
  - Hospital Universitario de Puerto Real, Cadiz, Andalusia
  - Institut Catalâ Oncologia-L'Hospitalet, L'Hospitalet de Llobregat, Barcelona [barcelona]
  - Hospital Universitario de Basurto, Bilbao, Bizkaia
  - Complejo Hospitalario Universitario de Vigo. Area Sanitaria de Vigo. Hospital Alvaro Cunqueiro, Vigo, Pontevedra, Cantabria Castilla Y LEON
  - Hospital General Universitario Morales Meseguer, Murcia, Comunidad de Murcia
  - Hospital San Jorge Huesca, Zaragoza, Huesca/ Aragon
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Hospital nuestra señora del prado de Toledo, Talavera de La Reina, Toledo, Madrid/castilla LA Mancha
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Clínico de Santiago de Compostela, Santiago de Compostela, Santiago de Compostela/cantabria
  - Hospital Universitario Virgen Del Rocio, Seville, Sevila
  - Hospital de Sagunto, Sagunto, Valencia, Valencia/madrid Castilla LA Mancha
  - Complejo Universitario de Albacete, Albacete
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Complejo Asistencial Universitario de Leon, León
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital de Sant Pau i Santa Tecla, Tarragona
  - Hospital Universitario Dr. Peset, Valencia
- Sweden (4):
  - Mälarsjukhuset, Eskilstuna, Södermanlands LÄN [se-04]
  - St Goran Hospital, Bromma
  - Örebro University Hospital, Örebro
  - Uppsala University Hospital, Uppsala
- Switzerland (2):
  - Kantonsspital Baden AG, Baden
  - Kantonsspital Baselland, Liestal
- United Kingdom (17):
  - Buckinghamshire Healthcare NHS Trust, Stoke Mandeville Hospital, Buckinghamshire, Buckinghamshire
  - Glan Clwyd Hospital, Rhyl, Denbighshire
  - Western General Hospital, Waterloo Place, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasglow, Glasglow City, Scotland
  - Ysbyty Gwynedd Hospital, Bangor, Gwynedd
  - Queen Elizabeth Hospital, Kings Lynn, Norfolk
  - Borders General Hospital, Roxburghshire, Scotland
  - Forth Valley Royal Hospital, Stirling, Scotland
  - Shrewsbury and Telford Hospital NHS Trust, Shrewsbury, Shropshire
  - Wrexham Maelor Hospital, Wrexham, Wales
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, WEST Yorkshire
  - Airedale NHS Foundation Trust, Keighley, WEST Yorkshire
  - Royal United Hospital Bath NHS Trust, Bath
  - Royal Blackburn Hospital, Blackburn
  - Royal Bournemouth Hospital, Bournemouth
  - Royal Cornwall Hospital, Cornwall
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481170